CLINICAL TRIAL: NCT06755580
Title: Comparison of Minimally Invasive Versus Open Spinopelvic Fixation for Unstable Sacral Fractures
Status: Completed | Type: Observational
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Hrin Tomas, MD, Principal investigator, F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Other Study IDs: 12/2024
Record Dates: First submitted 2024-12-20; First posted 2025-01-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Sacral Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients operated with open spinopelvic fixation: patients with vertically unstable high-energy sacral fracture operated with traditionally open spinopelvic fixation
  Interventions: Procedure: spinopelvic fixation
- patients operated with minimally invasive spinopelvic fixation.: patients with vertically unstable high-energy sacral fracture operated with minimally invasive spinopelvic fixation
  Interventions: Procedure: spinopelvic fixation

INTERVENTIONS:
Procedure: spinopelvic fixation — open and minimally invasive spinopelvic fixation for unstable or dislocated high-energy sacral fractures

SUMMARY:
The aim of this retrospective study is to evaluate patients with vertically unstable high-energy sacral fracture operated on at our institution with spinopelvic fixation, to compare the traditionally open method of fixation with the minimally invasive fixation. The aim of the research is to determine whether minimally invasive surgical techniques can achieve comparable fracture reduction and functional outcome as open surgical approaches. Another aim is to determine whether the minimally invasive surgical procedure leads to shorter patient hospitalization, lower perioperative blood loss, and lower postoperative complications.

DETAILED DESCRIPTION:
This retrospective study included 51 patients with vertically unstable sacral fracture operated at our institution with open or minimally invasive spinopelvic fixation over a period of 11 years (2014-2024). The patients were divided into two groups. One group of patients underwent open spinopelvic fixation, the other group underwent minimally invasive spinopelvic fixation. Each patient underwent a CT scan before and after surgery. The degree of fracture dislocation and reduction was measured in three planes at each examination. The degree of reduction was divided into four groups according to residual dislocation. In the perioperative period, blood loss, the length of the surgical procedure from the first incision to the suture of the wounds, and radiation exposure were monitored. Intraoperative blood loss was calculated from the waste in the surgical suction system. Functional outcome was assessed one year after surgery. A standardized questionnaire according to the Majeed score was used to assess functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* patient with high energy vertically unstable sacral fracture
* patients operated with open or minimally invasive spinopelvic fixation
* patients followed up for at least one year

Exclusion Criteria:

* patients with low-energy osteoporotic fractures of the sacrum
* patients with insufficiency fractures of the sacrum
* patients operated on using a method other than spinopelvic fixation
* patients who were not followed up for at least one year after surgery

Ages: 16 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients operated at our institution
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
pelvic ring symmetry | up to 1 year
  position of fracture fragments before and after surgery measured in three planes on CT scan
invasiveness of the surgical procedure | in perioperative period
  The invasiveness of the surgical procedure was measured based on perioperative blood loss. Perioperative blood loss was calculated from the waste in the surgical suction system (mililiters)
length of the surgical procedure | in perioperative period
  length of the surgical procedure from the first incision to the suture of the wounds
radiation exposure of the patient during surgical procedure | in perioperative period
  radiation exposure of a patient during a surgical procedure measured by the X-ray machine used during the operation (microgray/m2)
Functional outcome after surgery based on a standardized questionnaire according to the Majeed score | one year after surgery
  One year after surgery, patients fill out a standardized questionnaire according to the Majeed scoring system. Majeed score is a pelvic injury-specific functional assessment that comprises seven items, including pain, work, sitting, sexual intercourse, standing, unaided gait, and walking distance, with a total score range of 0 (worst outcome) to100 (best outcome), in order of decreasing disability.
complications | 1 year
  During the observation period, postoperative complications such as wound infection, loosening of osteosynthetic material, loss of reduction, nonunion, and newly developed neurological deficit will be recorded in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hrin, MD, Principal Investigator — F.D. Roosevelt Teaching Hospital with Policlinic
Locations (1):
- F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
plan to share all collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: starting in January 2025
Access Criteria: Data will be shared with medical journals for the purpose of publishing , with Slovak Medical University and with Slovak Medical Library for the purpose of clinical study report